CLINICAL TRIAL: NCT05982561
Title: Clinical Evaluation of BCDx for Monitoring of Recurrence in Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Type: Observational
Sponsor: Early is Good Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EIG 2023-02
Record Dates: First submitted 2023-07-27; First posted 2023-08-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
BCDx is a urine-based multi-omic assay for early cancer recurrence detection in patients with a history of bladder cancer. This prospective, blinded study evaluates its efficacy in detecting recurrent NMIBC, offering a noninvasive monitoring solution.

DETAILED DESCRIPTION:
BCDx is a urine-based multi-omic/multiplex molecular assay offers a promising solution for detecting cancer recurrence. It is intended for use as a noninvasive method for monitoring for tumor recurrence in conjunction with cystoscopy inpatients previously diagnosed with bladder cancer. This is a, multicenter, prospective, blinded study to evaluate the efficacy (sensitivity and specificity) of a novel multi-omics test for the detection of recurrent NMIBC in patients with a history of bladder cancer undergoing surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 Years and older
* Patients who have been diagnosed with incident or recurrent NMIBC within the past 2 years and undergoing standard of care/routine monitoring cystoscopy.
* Patients who are able to provide legally effective informed consent.
* Patients who are able to provide minimum 30mL of voided urine.

Exclusion Criteria:

* Patients planning to undergo radical cystectomy or chemotherapy-radiation for Urothelial Cell Carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cystoscopic surveillance for non-muscle invasive bladder cancer (NMIBC) follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) of BCDx (the proportion of negatives that are correctly identified as such by the gold standard) | Participants' urine samples will be collected before cystoscopy and analyzed using the BCDx test within 6 months to establish its overall performance characteristics.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arkansas Urology Research Center, Little Rock, Arkansas
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University, St Louis, Missouri